CLINICAL TRIAL: NCT04099641
Title: A Phase 2, Multicenter Open-label, Non-randomized Study of Bavituximab Plus Pembrolizumab in Patients With Advanced Gastric or Gastroesophageal Cancer Who Have Progressed on or After at Least One Prior Standard Therapy
Brief Title: An Open Label Study of Bavituximab and Pembrolizumab in Advanced Gastric and GEJ Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OncXerna Theraputics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCG100; 2019-000949-13 (EudraCT Number); KEYNOTE PN978 (Other: Merck)
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Gastric Cancer; GastroEsophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — bavituximab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- bavituximab and pembrolizumab (Experimental): Bavituximab 3mg/kg IV weekly in combination with pembrolizumab 200mg IV given once every 3 weeks
  Interventions: Drug: Bavituximab; Drug: Pembrolizumab Injection

INTERVENTIONS:
Drug: Bavituximab — Bavituximab IV infusion
Drug: Pembrolizumab Injection — Pembrolizumab IV Infusion
  Other Names: Keytruda

SUMMARY:
This study evaluates the combination of bavituximab and pembrolizumab in the treatment of gastric and gastroesphogeal cancer. All patients will receive both bavituximab, a drug that is not yet approved by the FDA, and pembrolizumab known as Keytruda.

There is no expanded access program available for the investigational agents per this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Men and women ≥ 18 years old; ≥ 20 years old in South Korea and Taiwan
* Unresectable metastatic or locally advanced gastric or GEJ adenocarcinoma
* Progressed on and/or after at least 1 prior regimen for metastatic disease or achieved stable disease or better in two consecutive scans to PD-1/PD-L1 inhibition alone or in combination with chemotherapy and relapsed
* Willing and able to provide fresh formalin-fixed paraffin-embedded tissue tumor sample
* Presence of at least one measurable lesion
* ECOG of 0 or 1
* Has adequate organ functions
* Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to start of study treatment.
* Women must not be breastfeeding.
* Women of childbearing potential , must agree to follow instructions for highly effective method(s) of contraception
* Males who are sexually active with women of childbearing potential must agree to follow instructions for highly effective method(s) of contraception
* Has adequate treatment washout period before start of study treatment

Exclusion Criteria:

* Received any form of anti-phosphatidylserine therapies
* Prior treatment with any checkpoint inhibitor or other therapies targeting T-cell control
* Known microsatellite instability-high (MSI-H) gastric or GEJ adenocarcinoma
* Medical history of myocardial infarction within 6 months before registration, symptomatic congestive heart failure (CHF) , troponin levels consistent with myocardial infarction, unstable angina, or serious cardiac arrhythmia
* Weight loss >10% over 2 months prior to first dose of study treatment
* History of pneumonitis that required steroids or has current pneumonitis
* Has known active CNS metastases/and or carcinomatous meningitis
* Known additional malignancy that is progressing or has required active treatment in within the past 3 years
* An active infection requiring systemic therapy
* Known human immunodeficiency virus (HIV) infection or known acute hepatitis B or C infection
* Unresolved toxicities from previous cancer treatments
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Active autoimmune disease or history of chronic recurrent autoimmune disease
* Severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
* History of infusion reactions to any component/excipient of bavituximab
* History of severe hypersensitivity reactions to mAbs.
* Systemic steroid therapy within 7 days prior to the first dose of study treatment
* Has received a live vaccine within 30 days prior to first dose of study drug.
* Prior organ transplantation including allogeneic or autologous stem-cell transplantation
* Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Receipt of treatment with immunotherapy, biological therapies, or therapeutic doses of hormonal therapies within 3 weeks of scheduled C1D1 dosing
* Known psychiatric, substance abuse disorder, or geographical travel limitations that would interfere with participant's ability to cooperate with the requirements of the study
* Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (9):
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Siteman Cancer Center - Washington University Medical Campus, St Louis, Missouri
  - White Plains Hospital - Center for Cancer Care, White Plains, New York
  - UC Health Office of Clinical Research, Cincinnati, Ohio
  - Cancer Treatment Centers of America at Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Sara Cannon Research Institute, Nashville, Tennessee
- South Korea (6):
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan District
- United Kingdom (2):
  - The Royal Marsden, London
  - Sarah Cannon Research Institute, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 25 centers located in 4 countries. A total of 107 participants were screened between 11 September 2019 and 03 June 2021, out of which 80 participants enrolled in the study.
Pre-assignment Details: A total of 80 participants received treatment: 61 participants had progressed on standard chemotherapy and were naïve to checkpoint inhibitor (CPI) therapy (CPI Naïve; Group 1) and 19 participants had achieved stable disease (SD) or better and then subsequently progressed following treatment with CPI either alone or in combination with chemotherapy (CPI Relapse; Group 2). Data are reported based on the date of 20 December 2021.
Groups:
- Group 1 (CPI Naïve): Group 1 participants had progressed on standard chemotherapy and were naïve to CPI therapy.
  Participants received bavituximab at 3 mg/kg on Days 1, 8, and 15 of a 3-week cycle through IV infusion. Participants received pembrolizumab at 200 mg on Day 1 of a 3-week cycle through IV infusion.
- Group 2 (CPI Relapse): Group 2 participants had achieved SD or better and then subsequently progressed following treatment with CPI either alone or in combination with chemotherapy.
  Participants received bavituximab at 3 mg/kg on Days 1, 8, and 15 of a 3-week cycle through IV infusion. Participants received pembrolizumab at 200 mg on Day 1 of a 3-week cycle through IV infusion.
Period: Overall Study
Arm/Group | Group 1 (CPI Naïve) | Group 2 (CPI Relapse)
Started | 61 | 19
Safety Population | 61 | 19
DLT-evaluable Population | 3 | 0
Efficacy Population | 61 | 19
Completed | 12 | 7
Not Completed | 49 | 12
Not completed — Death | 46 | 12
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety and efficacy populations included all participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (CPI Naïve) | Group 2 (CPI Relapse) | Total
Number analyzed (Participants) | 61 | 19 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (12.82) | 61.2 (11.68) | 60.4 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 4 | 20
  Male | 45 | 15 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 55 | 16 | 71
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 33 | 12 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 21 | 4 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 21 | 12 | 33
  United States | 27 | 4 | 31
  Taiwan | 11 | 0 | 11
  United Kingdom | 2 | 3 | 5
Central PD-L1 Combined Positive Score [Count of Participants; unit: Participants] — A combined positive score (CPS) was assessed for each FFPE-tumor specimen and defined by the number of PD-L 1 staining cells (tumor cells, lymphocytes, macrophages) divided by total number of tumor cells evaluated, multiplied by 100. The specimen should be considered to have PD-L 1 expression if CPS >=1 . The tumor cells are scored based on partial or complete membrane staining, which can be weak to strong in intensity (>=1 +). Staining in the immune cells (lymphocytes and macrophages) must also be >=1+.
  Participants
    <1 | 17 | 7 | 24
    ≥1 and <10 | 22 | 4 | 26
    ≥10 | 18 | 5 | 23
    Missing | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAE)
Description: Incidence of TEAEs graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0, including changes in clinical laboratory parameters. TEAEs: any AE that emerged on or after first dose, and within 30 days of the last dose.
Time Frame: From first dose through 30 days after last dose. Maximum exposure: 567 days.
Population: Analysis was performed on the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (CPI Naïve) | Group 2 (CPI Relapse)
Number analyzed (Participants) | 61 | 19
Participants | 61 | 19

2. Primary Outcome: Severity of Treatment Emergent Adverse Events (TEAE)
Description: Severity of TEAEs graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0, including changes in clinical laboratory parameters. TEAEs: any AE that emerged on or after first dose, and within 30 days of the last dose.
Time Frame: From first dose through 30 days after last dose. Maximum exposure: 567 days.
Population: Analysis was performed on the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (CPI Naïve) | Group 2 (CPI Relapse)
Number analyzed (Participants) | 61 | 19
Participants
  At least one Grade 1 TEAE | 3 | 4
  At least one Grade 2 TEAE | 19 | 2
  At least one Grade 3 TEAE | 21 | 8
  At least one Grade 4 TEAE | 1 | 0
  At least one Grade 5 TEAE | 17 | 5

3. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was based on RECIST version 1.1 criteria for target lesions, where a patient may achieve as best overall response (BOR) either complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD). CR was defined as the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline summary of diameters. ORR is calculated as the number of patients achieving a CR or PR (objective response) divided by the number of efficacy patients.
Time Frame: From date of first dose until the date of CR, PR, first documented progression or date of death from any cause, whichever came first. Maximum exposure: 567 days.
Population: The efficacy population include all participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (CPI Naïve) | Group 2 (CPI Relapse)
Number analyzed (Participants) | 61 | 19
Participants
  Complete Response | 2 | 0
  Partial Response | 6 | 1
  Stable Disease | 16 | 9
  Progressive Disease | 31 | 8
  Not Evaluable | 6 | 1

ADVERSE EVENTS:
Time Frame: From first dose through 30 days after last dose of study drug. Maximum exposure: 567 days.
Description: Safety population included all enrolled participants who received at least 1 dose of study drug, regardless of their eligibility for the study.
Arm/Group | Group 1 (CPI Naïve) | Group 2 (CPI Relapse)
All-Cause Mortality (participants affected / at risk) | 46/61 | 12/19
Serious Adverse Events (participants affected / at risk) | 29/61 | 10/19
Other Adverse Events (participants affected / at risk) | 61/61 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (CPI Naïve) (N=61) | Group 2 (CPI Relapse) (N=19)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 1
Disease progression (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Biliary tract infection (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Malignant urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (CPI Naïve) (N=61) | Group 2 (CPI Relapse) (N=19)
Anaemia (Blood and lymphatic system disorders) | 14 | 3
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 7 | 0
Constipation (Gastrointestinal disorders) | 16 | 9
Nausea (Gastrointestinal disorders) | 18 | 5
Diarrhoea (Gastrointestinal disorders) | 16 | 5
Vomiting (Gastrointestinal disorders) | 15 | 3
Abdominal pain (Gastrointestinal disorders) | 13 | 4
Abdominal pain upper (Gastrointestinal disorders) | 8 | 2
Abdominal distention (Gastrointestinal disorders) | 6 | 2
Ascites (Gastrointestinal disorders) | 5 | 3
Dysphagia (Gastrointestinal disorders) | 5 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 20 | 6
Oedema peripheral (General disorders) | 10 | 3
Pyrexia (General disorders) | 9 | 2
Asthenia (General disorders) | 6 | 1
Generalized oedema (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Swelling (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 1
Sepsis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 0 | 1
Emphysematous cholecystitis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Weight decreased (Investigations) | 10 | 3
Aspartate aminotransferase increased (Investigations) | 8 | 2
Alanine aminotransferase increased (Investigations) | 8 | 1
Blood alkaline phosphatase increased (Investigations) | 4 | 2
Blood bilirubin increased (Investigations) | 2 | 2
Blood creatinine increased (Investigations) | 4 | 0
Blood cholesterol increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1
Liver function test increased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 21 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 3
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 7 | 4
Dizziness (Nervous system disorders) | 9 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 2
Depression (Psychiatric disorders) | 5 | 0
Dysuria (Renal and urinary disorders) | 3 | 2
Obstructive nephropathy (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2
Hypertension (Vascular disorders) | 7 | 1
Hypotension (Vascular disorders) | 3 | 1
Vision blurred (Eye disorders) | 2 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 1
Chills (General disorders) | 8 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT04099641/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT04099641/SAP_001.pdf